CLINICAL TRIAL: NCT00697450
Title: Observational Study Evaluating the Body Weight Progress During the Treatment With Insulin Detemir (Levemir®) in Type 2 Patients, Previously Treated With Other Basal Insulins
Brief Title: Observational Study on the Weight Effect of Insulin Detemir (Levemir®) in Type 2 Diabetics
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3560
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose, frequency of dosing, dose titration to be prescribed by the physician as a result of a normal clinical evaluation

SUMMARY:
This study is conducted in Europe. Observational study evaluating the body weight progress during the treatment with insulin detemir (Levemir®) in Type 2 patients, previously treated with other basal insulins

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Current treatment with insulin NPH or glargine
* The selection of the subjects will be at the discretion of the individual physician

Exclusion Criteria:

* Current treatment with insulin detemir
* Previous enrolment in this study
* Hypersensitivity to insulin detemir or to any of the excipients.
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetics
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Weight effect | 12 months prior to and 12 months after detemir treatment.

SECONDARY OUTCOMES:
Improvement in FPG levels | 12 months prior and 12 months after detemir treatment
Improvement in HbA1c levels | 12 months prior and 12 months after detemir treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Prague, Czechia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com